CLINICAL TRIAL: NCT04808050
Title: A Multicountry, Multicentre, Non-interventional, Retrospective Study to Determine the Real-world Treatment Patterns and Associated Outcomes in Patients With Resectable Early-stage (IA to IIIB) Non-small Cell Lung Cancer
Brief Title: Real-world Treatment Patterns and Associated Outcomes in Patients With Resectable Early-stage Non-small Cell Lung Cancer
Acronym: THASSOS-INTL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00169
Record Dates: First submitted 2021-02-22; First posted 2021-03-19 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Resectable Early-stage (IA to IIIB)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, multi-country, multicentre, retrospective study designed to determine the treatment patterns and associated survival rate in patients with primary stage IA to IIIB resectable NSCLC diagnosed between 01 January 2013 and 31 December 2017 and followed until at least 31 December 2020 The main objective of this study is to describe the treatment patterns and determine their associated 3-year survival rate according to clinical and pathologic staging in patients with resectable early-stage (IA to IIIB as per AJCC seventh edition) NSCLC.

DETAILED DESCRIPTION:
This is a non-interventional, multi-country, multicentre, retrospective study designed to determine the treatment patterns and associated survival rate in patients with primary stage IA to IIIB resectable NSCLC diagnosed between 01 January 2013 and 31 December 2017 and followed until at least 31 December 2020. This study will also determine the prevalence of EGFR mutations and PD-L1 expression, and the clinical outcomes as per the treatment patterns and clinico-pathological staging. Data will be collected retrospectively from the patients' medical records from the date of initial diagnosis of early-stage NSCLC (index date) to the end of follow up ie, until death, the last medical record entry, or date of data extraction, whichever is the earliest. The data on treatment modalities, sociodemographic, clinico-pathological characteristics, and exposure and outcome variables (ie, medical and treatment history, disease staging, biomarker assessments, radiological findings, concomitant medications, survival), factor(s) for prescribing neo-adjuvant and/or adjuvant treatment and reason(s) for discontinuation will be extracted from patients' medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female and male patients aged ≥18 years or 'adults' according to age of majority as defined by the local regulations on index date
2. Patient or next of kin/legal representative (for deceased patients at study entry, unless a waiver is granted) willing and able to provide written or electronic informed consent according to the local regulations, where applicable
3. Patients diagnosed with primary stage IA to IIIB NSCLC as per seventh edition AJCC whose tumour was deemed resectable between 01 January 2013 and 31 December 2017 and followed up until at least 31 December 2020, as per the medical records with availability of at least 12 months of follow-up data from the index date (date of diagnosis of early-stage [IA to stage IIIB] resectable NSCLC), unless patient died within 12 months of diagnosis.

Exclusion Criteria:

1. Patients with a concomitant cancer at the time of diagnosis of NSCLC, except for nonmetastatic nonmelanoma skin cancers, or in situ or benign neoplasms; a cancer will be considered concomitant if it occurs within 5 years of NSCLC diagnosis
2. Patients diagnosed with stage IV NSCLC
3. Histology of the tumour is small cell lung cancer, neuroendocrine in origin, or a mixed histologic type with small cell and non-small cell lung cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with primary stage IA to IIIB NSCLC between 01 January 2013 and 31 December 2017 and followed up until at least 31 December 2020.
Sampling Method: Probability Sample
Enrollment: 748 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients per treatment modalities | 3 Years
  Proportion of patients, overall and as per clinical and pathologic staging (seventh edition of the tumour, nodes, metastases [TNM] classification for lung cancer [AJCC]) who underwent treatment Surgery only, Neo-adjuvant therapy (chemo+/-radiotherapy) only, Adjuvant therapy (chemo+/-radiotherapy) only or Neo-adjuvant and adjuvant therapies modalities
Duration of treatment | 3 years
  Duration of treatment for each treatment regimen in neo-adjuvant and adjuvant treatment settings, dose of each agent, and reason(s) for stopping treatment in each setting
Survival rate | 3 Years
  Survival rate (overall, and as per clinical and pathologic staging) defined as percentage of patients, confirmed to be alive at 3 years from the index date.

SECONDARY OUTCOMES:
Demographic characteristics | 3 Years
  Demographic overall and as per treatment modalities ; underwent treatment Surgery only, Neo-adjuvant therapy (chemo+/-radiotherapy) only, Adjuvant therapy (chemo+/-radiotherapy) only or Neo-adjuvant and adjuvant therapies modalities): age, gender, ethnicity, body mass index, smoking status, geographical location
Eastern Cooperative Oncology performance status Group characteristics | 3 Years
  Proportion and classification of Eastern Cooperative Oncology Group (ECOG) performance status Clinical-pathological characteristics overall and as per treatment modalities ; underwent treatment Surgery only, Neo-adjuvant therapy (chemo+/-radiotherapy) only, Adjuvant therapy (chemo+/-radiotherapy) only or Neo-adjuvant and adjuvant therapies modalities
Histological type | 3 Yewars
  Proportion of Histological type (adenocarcinoma, adenosquamous carcinoma, bronchioalveolar carcinoma, large-cell carcinoma, and NSCLC not otherwise specified)
Clinical-pathological Tumor stage | 3 Years
  Tumor Staging as per seventh edition AJCC (IA, IB, IIA, IIB, IIIA, IIIB) with lymph node metastasis status (N0, N1, and N2)
TNM staging at index diagnosis | 1 Month
  TNM staging at index diagnosis
Genetic alterations | 3 Years
  Other genetic alterations(anaplastic lymphoma kinase [ALK], Kirsten rat sarcoma viral oncogene [KRAS], B-Raf proto-oncogene [BRAF], rearranged during transfection [RET], mesenchymal-to-epithelial transition factor [MET], human epidermal growth factor receptor 2 [HER2], ROS proto-oncogene 1 receptor tyrosine kinase [ROS1], and tumour protein 53 [TP53]
Survival rates at pre-defined landmark timepoints (other than 3-year) | 1 Years
  Survival rates at pre-defined landmark timepoints (other than 3-year) for each of the treatment modality; ho underwent treatment Surgery only, Neo-adjuvant therapy (chemo+/-radiotherapy) only, Adjuvant therapy (chemo+/-radiotherapy) only or Neo-adjuvant and adjuvant therapies
Prevalence of EGFR mutations | 3 Years
  Proportion of patients with EGFR mutation-positive status
Prevalence of PD-L1 expression | 3 Years
  Proportion of patients with PD-L1 positivity at various cut-off points (<1%, ≥1% to <25%, ≥25% to <50%, and ≥50%)

OTHER OUTCOMES:
Effectiveness outcomes rwDFS defined as time from the date of surgery to recurrence or death | 3 Years
  Effectiveness outcomes will be determined for each treatment modality as; rwDFS defined as time from the date of surgery to recurrence or death due to any cause; rwDFS rate at predefined landmark timepoints (overall, per clinical, and pathologic staging) for evaluation of primary treatment
Effectiveness outcomes rwEFS rate at predefined landmark timepoints | 3 Years
  Effectiveness outcomes will be determined for each treatment modality as; rwEFS rate at predefined landmark timepoints (overall, per clinical and pathologic staging) for evaluation of primary treatment
Effectiveness outcomes rwPFS defined as time from local or distant relapse to disease progression or death | 3 Years
  Effectiveness outcomes will be determined for each treatment modality as; rwPFS defined as time from local or distant relapse to disease progression or death due to any cause for evaluation of subsequent treatment ie, first, second, and third LOTsa

CONTACTS AND LOCATIONS:
Locations (23):
- Australia (3):
  - Research Site, Sydney, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Perth, Western Australia
- Egypt (3):
  - Research Site, Alexandria
  - Research Site, Cairo
  - Research Site, Sohag
- Research Site, Hong Kong, Hong Kong
- India (7):
  - Research Site, Howrah, Kolkata, India
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Faridabad
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, New Delhi
- Research Site, Kuwait City, Kuwait
- Turkey (Türkiye) (7):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Diyarbakır
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Samsun
- Research Site, Alain, United Arab Emirates, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  URL:
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00169&attachmentIdentifier=a46a5a9f-c86c-4048-a611-8c7fd9910625&fileName=THASSOS_D133FR00169_CSR_1.0__31_Jan_2023_Redacted.pdf&versionIdentifier=